CLINICAL TRIAL: NCT04342156
Title: Safety And Efficacy Of Hydroxychloroquine For At Risk Population (SHARP) Against COVID-19- A Cluster Randomized Controlled Trial (SHARP COVID-19 RCT)
Brief Title: Safety And Efficacy Of Hydroxychloroquine For At Risk Population (SHARP) Against COVID-19
Acronym: SHARP COVID-19
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The number of patients with COVID-19 in Singapore was coming down for the community and the concerns about the potential side effects particularly when the baseline ECG and serum electrolytes was not proposed.
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: National Center for Infectious Diseases (Other Government); Singapore Clinical Research Institute (Other); Singapore Eye Research Institute (Other); Saw Swee Hock School of Public Health (Unknown); Duke-NUS Graduate Medical School (Other); Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/00402
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Infection; Hydroxychloroquine Adverse Reaction
Keywords: Post Exposure Prophylaxis (PEP); Hydroxychloroquine; Singapore; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Treatment arm will be given Hydroxychloroquine sulfate. Dose: 800 milligrams (mg) (4 pills of 200mg) in two divided doses on day 1 followed by 400mg (2 pills of 200mg) in two divided doses on day 2, 3,4, 5.
  Mode of administration: Oral pills of 200mg of HCQ; Supply: The total supply of all the pills (12 pills of 200mg per subject in the study group) will be given to the recruited subject from day 1.
  Interventions: Drug: Hydroxychloroquine Sulfate 200 milligram (mg) Tab
- Standard Preventive Measures (Other): No intervention. Standard recommended preventive measures by the ministry of health.
  Interventions: Drug: Hydroxychloroquine Sulfate 200 milligram (mg) Tab

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 200 milligram (mg) Tab — Oral tablet of Hydroxychloroquine sulfate

SUMMARY:
The Coronavirus Disease 2019 (COVID-19) pandemic has placed tremendous stress on the global economy since its outbreak in December 2019. Currently, with nearly 1.3 million confirmed cases, there is still no effective way to contain the disease. The transmission of COVID-19 occurs via direct (prolonged close interaction, within 2 meters for more than 30 minutes) and indirect (fomites) contacts. Locally, the risk of COVID-19 infection in household contacts of confirmed cases is about 4%. These at-risk individuals are identified through contact tracing and infectious may be preventable using post-exposure-prophylaxis (PEP). However, there has yet to be a single effective, safe, and affordable pharmacological agent with such capabilities. Hydroxychloroquine (HCQ) is a cheap anti-malarial and immunomodulatory agent which may potentially be used as PEP against COVID-19. HCQ is capable of blocking the invasion and intracellular replication of the virus. Existing studies have reported efficacy of HCQ in treating COVID-19, with reduced time to clinical recovery and few reports of patients suffering from significant side effects. However, existing studies are largely limited by their small sample sizes. Furthermore, there has yet to be a published trial on HCQ's role in PEP. This cluster randomized trial will evaluate the safety and efficacy of oral HCQ PEP, taken over for 5 days, in reducing the number of infected household contacts of confirmed COVID-19 patients under home quarantine. Comparison will be made between HCQ PEP (treatment group) and no treatment (control group). Subjects will be followed up over a course of 28 days, with daily symptom monitoring conducted over phone calls. Positive outcomes from this study will provide a means for us to battle the COVID-19 pandemic.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18 to 80 years.
2. History of close contact or exposure to positive COVID-19 cases in the same household.
3. Absence of symptoms resembling COVID-19 (e.g., fever and acute respiratory or gastrointestinal symptoms) for two weeks prior to enrolment for the study.
4. Able to give informed consent or in case of <21 and>/=18 years old subject, parents able to give consent for those individuals. In the event the household is unable to read or sign/date the ICF, an impartial witness to be present to ascertain the information, comprehension and voluntariness. The impartial witness must be able to read the informed consent form (ICF).
5. Able to comply with study procedures and follow-up
6. Singapore citizen, permanent resident or long-term pass-holder.

Exclusion Criteria:

1. Person diagnosed with COVID-19 infection.
2. Pregnant at the time of screening or breastfeeding.
3. Known allergy or hypersensitivity to HCQ or other aminoquinoline compounds.
4. Already on HCQ for different indications (e.g., rheumatological diseases, malaria prophylaxis)
5. Diagnosis of other systemic viral or bacterial infection.
6. Use of systemic immunosuppressant agents within 90 days of enrollment (e.g., corticosteroids and immunomodulatory therapy)
7. History of immunocompromised state.
8. History of psychiatric illness.
9. History of psoriasis or porphyria.
10. History of cardiac disease.
11. Other major comorbidities that contraindicate the use of HCQ: i. Hematologic malignancy, ii. Stage 4-5 chronic kidney disease or end-stage renal failure, iii. history of ventricular arrhythmias, iv. current use of drugs that prolong the QT interval
12. History of severe skin reactions such as Stevens-Johnson syndrome and toxic epidermal necrolysis.
13. Bradycardia <50beats/min.
14. Uncorrected hypokalemia
15. Uncorrected hypomagnesemia.
16. Unwillingness to practice acceptable methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) while on study and for at least 30 days after last dose.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
positive serology or reverse transcriptase (RT-PCR) for COVID-19 up until day 28. | Until day 28
  COVID-19 infection

SECONDARY OUTCOMES:
Positive serology at day 28. | 28 days
  Serology
Symptoms of COVID-19. | Until day 28
  COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Rupesh Agrawal, MD, Principal Investigator — Tan Tock Seng Hospital

IPD SHARING:
Plan to Share IPD: No